CLINICAL TRIAL: NCT04012788
Title: The Effectiveness of a Synbiotic Mixture (Inulin, Lactobacillus Rhamnosus (LGG®), Lactobacillus Acidophilus (LA-5®), Lactobacillus Paracasei, and Bifidobacterium Lactis (BB-12®)), on Decreasing Recurrence of Clostridium Difficile Associated Diarrhea- a , Randomized, Placebo-controlled Study With 4 Weeks Intervention
Brief Title: CDI Synbiotic Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Andreas Munk Petersen, MD, Cosultant, PhD, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H-18041764
Record Dates: First submitted 2019-04-05; First posted 2019-07-09 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Clostridium Difficile Infection
Keywords: probiotics; prebiotics; synbiotics
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- probiotic arm (Active Comparator): inulin, 15 g Lactobacillus rhamnosus (LGG®) Lactobacillus acidophilus (LA-5®) Lactobacillus paracasei (L. casei 431®) Bifidobacterium lactis (BB-12®), Total cell counts 150 billion/day
  Interventions: Dietary Supplement: Synbiotic mixture
- placebo arm (Placebo Comparator): placebo powder, 15 g
  Interventions: Other: Placebo comparator

INTERVENTIONS:
Dietary Supplement: Synbiotic mixture — A synbiotic mixture consisting of four probiotic strains and inulin (a prebiotic)
  Arms: probiotic arm
Other: Placebo comparator — Placebo powder
  Arms: placebo arm

SUMMARY:
The investigators hypothesize that treatment with a synbiotic mixture consisting of inulin Lactobacillus rhamnosus (LGG®), Lactobacillus acidophilus (LA-5®), Lactobacillus paracasei (L. casei 431®) and Bifidobacterium lactis (BB-12®) can reduce the number of C. difficile recurrences significantly.

DETAILED DESCRIPTION:
Probiotics have been tested for their efficacy in preventing infection with C. difficile after antibiotic exposure. Some of the most effective probiotics tested Lactobacillus rhamnosus (LGG®), Lactobacillus acidophilus (LA-5®), Lactobacillus paracasei (L. casei 431®) and Bifidobacterium lactis (BB-12®). However, most studies have focused on prevention of the first incidence of C. difficile infection rather than prevention of re-infection with C. difficile. Recurrence rates of C. difficile infection (CDI) among hospitalized patients are 15-25% - either as relapses caused by the original organism or re-infection following treatment. The potential of probiotics in preventing re-infection is less studied in these patients. Further, prebiotics which are carbohydrates only metabolized by beneficial bacteria have gained much attention the recent years for their health benefits through stimulating growth of specific types of bacteria in the gut, and recent data from mouse studies show that the prebiotic inulin can eliminate C. difficile growth, but the use of prebiotics in relation to C. difficile elimination has yet to be proven in humans. The investigators hypothesize that treatment with a synbiotic mixture consisting of inulin Lactobacillus rhamnosus (LGG®), Lactobacillus acidophilus (LA-5®), Lactobacillus paracasei (L. casei 431®) and Bifidobacterium lactis (BB-12®) can reduce the number of C. difficile recurrences significantly.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with primary CDI
* Treatment with Vancomycin
* Subjects over 18 years of age
* Signed informed consent

Exclusion Criteria:

1. Chemotherapy within two months and an absolute neutrophil count of < 1000 neutrophiles/mm3
2. Acute leukemia
3. Serious immunodeficiency
4. Pancreatitis
5. Planned or recent intraabdominal operation within a time window of 14 days
6. Terminal disease with expected survival time < 3 month
7. Probiotic consumption within two weeks prior enrollment
8. Pregnant or lactating women
9. A history of inflammatory or irritable bowel disease
10. Colectomy and cirrhosis
11. Septicemia
12. Toxic megacolon

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-07 (Estimated); Primary Completion 2020-05-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Reduced recurrence of C. difficile-associated diarrhoea (CDAD) after 8 weeks | 1 year
  telephone questionnaire with patient at end of trial as well as examination of each patient's medical record

SECONDARY OUTCOMES:
toxin A and B levels measured by qPCR | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Andreas M Petersen, Principal Investigator — Gastrounit, Hvidovre Hospital
Locations (1):
- Hvidovre Hospital, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: No